CLINICAL TRIAL: NCT02879266
Title: Phase I Evaluation of the Safety and Immunogenicity of an Investigational Tetravalent Dengue Vaccine (TetraVax-DV) TV005 in Flavivirus-Naïve Adults 50 - 70 Years of Age
Brief Title: Evaluating the Safety and Immunogenicity of a Tetravalent Dengue Vaccine (TetraVax-DV) TV005 in Flavivirus-Naive Adults 50 to 70 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 310
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Dengue
Keywords: Dengue Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TetraVax-DV TV005 (Experimental): Participants will receive a subcutaneous injection of TetraVax-DV TV005 at study entry (Day 0).
  Interventions: Biological: TetraVax-DV TV005
- Placebo (Placebo Comparator): Participants will receive a subcutaneous injection of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TetraVax-DV TV005 — Contains 10^3 plaque-forming units (PFUs) of rDEN1Δ30, 10^4 PFUs of rDEN2/4Δ30(ME), 10^3 PFUs of rDEN3Δ30/31-7164, and 10^3 PFUs of rDEN4Δ30; administered by subcutaneous injection in the deltoid region of the upper arm
  Other Names: TV005
  Arms: TetraVax-DV TV005
Biological: Placebo — Administered by subcutaneous injection in the deltoid region of the upper arm
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and immunogenicity of a tetravalent dengue vaccine TetraVax-DV TV005 in adults 50 to 70 years of age with no history of previous flavivirus infection.

DETAILED DESCRIPTION:
Dengue viruses (DENV) are widespread in most tropical and subtropical regions of the world. There are four serotypes of dengue virus (DENV-1, DENV-2, DENV-3, and DENV-4); each can cause dengue infection. Infection with dengue viruses can range from mild illness to life-threatening disease. TetraVax-DV TV005 (also referred to as TV005) is a live attenuated recombinant tetravalent dengue virus vaccine developed to protect against all four dengue virus serotypes. The purpose of this study is to evaluate the safety and immunogenicity of TV005 in adults 50 to 70 years of age with no history of previous flavivirus infection.

Participants will be randomly assigned to receive a subcutaneous injection of either TV005 or placebo at study entry (Day 0). After receiving the injection, participants will record their temperature 3 times a day through Day 16. Additional study visits will occur on Days 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, and 180. Visits will include a physical examination and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult flavivirus-naive male or non-pregnant females 50 - 70 years of age, inclusive
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-vaccination
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females only: Female subjects of childbearing potential willing to use effective contraception. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (6 months or longer since last sexual encounter). All female subjects will be considered having childbearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Currently pregnant, as determined by positive beta-human choriogonadotropin (HCG) test; or breastfeeding (females only)
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC) or alanine aminotransferase (ALT), as defined in this protocol
* Serum creatinine level above the laboratory-defined upper limit of normal
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications)
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 21 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* History and/or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination
* Definite plan to travel to a dengue-endemic area during the study
* Refusal to allow storage of specimens for future research

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Frequency of TV005-related adverse events (AEs) | Measured through Day 180
  AEs classified by both severity and seriousness, through active and passive surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland, United States